CLINICAL TRIAL: NCT03090191
Title: A PHASE 3, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF A CLOSTRIDIUM DIFFICILE VACCINE IN ADULTS 50 YEARS OF AGE AND OLDER
Brief Title: Clostridium Difficile Vaccine Efficacy Trial
Acronym: Clover
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B5091007; 2016-003866-14 (EudraCT Number); CLOVER (Other: Alias Study Number)
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clostridium difficile vaccine (Experimental)
  Interventions: Biological: Clostridium difficile vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Clostridium difficile vaccine — Toxoid-based Clostridium difficile vaccine
  Arms: Clostridium difficile vaccine
Biological: Placebo — Normal saline solution (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
The Clover trial is evaluating an investigational vaccine that may help to prevent Clostridium difficile infection. Participants in the study are adults 50 years of age and older, who are at risk of developing Clostridium difficile infection. The study will assess whether the vaccine prevents the disease, and whether it is safe and well tolerated.

Each subject will receive 3 doses of Clostridium difficile vaccine or placebo and be followed for up to 3 years after vaccination for potential Clostridium difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Willing and able to comply with study procedures.
* Subjects with an increased risk of future contact with healthcare systems or subjects who have received systemic antibiotics in the previous 12 weeks.
* Ability to be contacted by telephone during study participation.
* Negative urine pregnancy test for female subjects of childbearing potential.

Exclusion Criteria:

* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s)/vaccine(s) within 28 days prior to study entry until 1 month after the third vaccination.
* Previous administration of an investigational C difficile vaccine or C difficile mAb therapy.
* Prior episode of CDI..
* Receipt of blood products or immunoglobulins within 6 months before enrollment.
* Subjects who may be unable to respond to vaccination due to:

  * Metastatic malignancy; or
  * End-stage renal disease; or
  * Any serious medical disorder likely to be fatal within the next 12 months; or
  * Congenital or acquired immunodeficiency; or
  * Receipt of high dose systemic corticosteroids for 14 days within 28 days of enrollment; or
  * Receipt of chronic systemic treatment with other known immunosuppressant medications, or radiotherapy, within 6 months of enrollment.
* Known infection with human immunodeficiency virus (HIV).
* Any bleeding disorder or anticoagulant therapy that would contraindicate intramuscular injection.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.
* Prior small- or large-bowel resection.
* Any condition or treatment resulting in frequent diarrhea.
* Other acute or chronic condition or abnormality that may increase the risk associated with study participation or IP administration or may interfere with interpretation of study results
* Pregnant or breastfeeding female subjects; male subjects and female subjects who are sexually active and at risk for pregnancy and will not/cannot use 2 methods of contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17535 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (426):
- United States (220):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Coastal Clinical Research, LLC, An AMR Company, Mobile, Alabama
  - The Pain Center of Arizona, Peoria, Arizona
  - Phoenix VA Health Care System, Phoenix, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Baptist Health Rehabilitation Institute, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - California Kidney Specialist, Covina, California
  - Usborne Family Medicine, Covina, California
  - Kaiser Permanente Daly City, Daly City, California
  - Premier Health Research Center, LLC, Downey, California
  - Paradigm Clinical Research Centers, Inc., La Mesa, California
  - VA Loma Linda Healthcare System Research Pharmacy, Loma Linda, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - Long Beach Clinical Trials, Long Beach, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Academic Medical Research Institute, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA CTRC Outpatient Unit, Los Angeles, California
  - VA Northern California Health Care System, Mather, California
  - Veterans Affairs Palo Alto Health Care System, Palo Alto, California
  - Covigilant Research, LLC, Rancho Mirage, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - VA Loma Linda Healthcare System Ambulatory Care System, Redlands, California
  - Covigilant Research LLC, Riverside, California
  - Kaiser Permanente Roseville, Roseville, California
  - One Community Health, Sacramento, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - CTSC Clinical Research Center, Sacramento, California
  - Lawrence J. Ellison Ambulatory Care Center, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente South Sacramento, Sacramento, California
  - Breakthrough Clinical Trials, San Bernardino, California
  - VA San Diego Healthcare System, San Diego, California
  - California Kidney Specialists, San Dimas, California
  - Kaiser Permanente San Jose, San Jose, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Alta California Medical Group, Simi Valley, California
  - Kaiser Permanente Walnut Creek, Walnut Creek, California
  - Clinical Trial Center University of Colorado Denver, School of Medicine, Aurora, Colorado
  - University of Colorado Clinical & Translational Research Center Clinic, Aurora, Colorado
  - University of Colorado Clinical & Translational Research Center Outpatient Clinic, Aurora, Colorado
  - University of Colorado Denver, School of Medicine, Aurora, Colorado
  - University of Colorado Department of AIP 2. Pharmacy Bulk Storage, Aurora, Colorado
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Florida Sleep Disorder Center of Brandon, Brandon, Florida
  - Teradan Clinical Trials, Brandon, Florida
  - Southeast Clinical Research, Chiefland, Florida
  - Innovative Research of West FL., Inc., Clearwater, Florida
  - Alliance for Multispecialty Reseach, LLC, Coral Gables, Florida
  - Omega Research Consultants, LLC, DeBary, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Malcom Randall VA Medical Center Investigational Drug Services, Gainesville, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions,Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Optimus U. Corp., Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Doctors Research Institute, Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - HMD Research LLC, Orlando, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Soma Medical Center, West Palm Beach, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Christie Clinic, LLC, Champaign, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Springfield Clinic Infectious Diseases, Springfield, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Infectious Disease of Indiana, PSC, Carmel, Indiana
  - St. Vincent Outpatient Treatment Center, Carmel, Indiana
  - Deaconess Clinic Mt. Pleasant, Evansville, Indiana
  - St. Vincent Hospital & Health Care Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - MOC Research, Mishawaka, Indiana
  - Meridian Clinical Research, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Central Kentucky Research Associates, LLC, Lexington, Kentucky
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - Barnum Medical Research Inc, Natchitoches, Louisiana
  - Ochsner Center for Primary Care and Wellness, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Luminis Health Anne Arundel Medical Center Infusion Center, Annapolis, Maryland
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Luminis Health Research Institute: Research Office, Annapolis, Maryland
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - ClinSite, LLC, Canton, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Revival Research Institute, LLC, Sterling Heights, Michigan
  - Mayo Clinic Rochester, Methodist Hospital Campus, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - MedPharmics, Gulfport, Mississippi
  - Center for Outpatient Health, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Center For Clinical Studies, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Bozeman Health Deaconess Hospital d/b/a Bozeman Health Clinical Research, Bozeman, Montana
  - Bozeman Health GI Clinic, Bozeman, Montana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Barrett Clinic, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - ID Care, Hillsborough, New Jersey
  - Amici Clinical Research, Raritan, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - Meridian Clinical Research LLC, Binghamton, New York
  - Meridian Clinical Research, LLC, Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Durham VAMC, Durham, North Carolina
  - Duke Early Phase Clinical Research, Durham, North Carolina
  - Duke University Hospital Investigational Drug Services (IDS) Pharmacy, Durham, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Waterway Primary Care LLC DBA Tabor City Family Medicine, Tabor City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Aultman Cardiology Clinical Trials, Canton, Ohio
  - Aultman Hospital, Canton, Ohio
  - UC Health Physicians Office Clifton, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - University Of Cincinnati-Internal Medicine Division of Digestive Diseases, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Remington-Davis, Incorporated, Columbus, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Great Lakes Medical Research LLC, Mentor, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Kaiser Permanente Center For Health Research, Portland, Oregon
  - Columbia Research Group, Inc., Portland, Oregon
  - VA Portland Healthcare System, Portland, Oregon
  - Lehigh Valley Health Network/Network Office of Research and Innovation, Allentown, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Westminster Family Medicine, Erie, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Uniontown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Medical Research South, LLC, Charleston, South Carolina
  - Main Street Physician's Care - Waterway, Little River, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - PMG Research,Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Synexus US, LP, Dallas, Texas
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Synexus US, dba Research Across America, Mesquite, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - South Texas Veterans Healthcare System, Audie L Murphy Hospital, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - Advanced Clinical Research/Gut Whisperer, Riverton, Utah
  - J. Lewis Research, Inc./Foothill Family Clinic, Salt Lake City, Utah
  - J Lewis Research, Incorporated, Salt Lake City, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC, Annandale, Virginia
  - Virginia Research Center LLC, Midlothian, Virginia
  - Salem VAMC, Salem, Virginia
  - Frandsen Family Medicine DBA Sound Medical Research, Port Orchard, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Universal Research Group, LLC, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Marshfield Medical Center - Marshfield, Marshfield, Wisconsin
- Argentina (5):
  - Hospital Aleman, C.a.b.a., Buenos Aires
  - Hospital Italiano de Buenos Aires, C.a.b.a., Buenos Aires
  - Centro Médico Dra. De Salvo, C.a.b.a., Buenos Aires
  - Sanatorio Británico S.A., Rosario, Santa Fe Province
  - Hospital Nuestra Senora de la Misericordia, Córdoba
- Australia (12):
  - Paratus Clinical Pty Ltd, Kanwal, New South Wales
  - Australian Clinical Research Network, Maroiubra, New South Wales
  - Maroubra Medical Centre, Maroubra, New South Wales
  - University Clinic Pharmacy, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Austrials Pty Ltd, Sherwood, Queensland
  - Mater Misericordiae Ltd & Mater Medical Research Institute Ltd, South Brisbane, Queensland
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - Australian Clinical Research Network, Maroubra
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
  - CHU de Liège - Domaine universitaire du Sart Tilman, Liège
- Bulgaria (17):
  - "MHAT- Dr. Hristo Stambolski" EOOD, Kazanlak
  - MHAT ''Sv.Ivan Rilski-Kozloduy'' EOOD; Internal Department, Kozloduy
  - MHAT "Sv. Nikolay Chudotvorets" EOOD, Lom
  - UMHAT "Dr. Georgi Stranski" EAD, Second Psychiatric Clinic of general psychiatry and dependence, Pleven
  - UMHAT "Sveti Georgi" EAD, Plovdiv
  - "Center for Mental Health - Ruse" EOOD, Rousse
  - SHATPPD Dr. Dimitar Gramatikov - Ruse EOOD, Rousse
  - ''Medical Center-1-Sevlievo'' EOOD, Sevlievo
  - MHAT -Silistra AD, Silistra
  - MC ''Tsaritsa Yoanna''EOOD, Sliven
  - MC 'Cardiohelp' EOOD, Sofia
  - "Acibadem City Clinic University Hospital" EOOD, Sofia
  - Acibadem City Clinic Tokuda Ead, Sofia
  - MHAT "Sveta Anna - Sofia" AD, Clinic of Internal Diseases, Sofia
  - "SHATPD-Troyan" EOOD, Troyan Municipality
  - MC Medica Plus OOD, Veliko Tarnovo
  - MHAT ''Sveta Petka" AD, Vidin
- Canada (12):
  - Vancouver Coastal Health Research Institution-clinical research unit-Diamond Health Care Centre, Vancouver, British Columbia
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - The Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Manna Research Inc. (Toronto), Toronto, Ontario
  - Intermed Groupe Santé, Chicoutimi, Quebec
  - Q & T Research Outaouais Inc., Gatineau, Quebec
  - Centre Integre de Sante et de Services Sociaux de la Monteregie- Center- Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Centre de recherche du CHU de Quebec-Universite Laval, Québec, Quebec
  - Centre de recherche Saint-Louis, Québec, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
  - Centre Integre Universitaire de Santé et de Services Sociaux de la Mauricie et du Centre du Québec, Trois-Rivières, Quebec
- Chile (5):
  - Psicomed Esudios Medicos, Antofagasta, Antofagasta
  - Centro de Investigacion Clínica del Sur, Temuco, IX Region de LA Araucania
  - Hospital Dr. Hernan Henriquez Aravena, Temuco, Región de la Araucanía
  - Biomedica Research Group, Santiago, Santiago Metropolitan
  - Fundacion Arriaran, Santiago, Santiago Metropolitan
- Colombia (10):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Fundacion Centro de Investigacion Clinica - CIC, Medellín, Antioquia
  - Instituto de Coloproctologia ICO, Medellín, Antioquia
  - Clinica de la Costa Ltda., Barranquilla, Atlántico
  - Asociación IPS Médicos Internistas de Caldas, Manizales, Caldas Department
  - Centro de Investigaciones - MedPlus Centro de Recuperación Integral S.A.S., Bogotá, D.C.
  - Fundación Cardiomet CEQUIN, Armenia, Quindío Department
  - Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A., Cali, Valle del Cauca Department
- Czechia (11):
  - Doktor Brno s.r.o., Brno, Czech
  - Ordinace vseobecneho praktickeho lekare, Benátky nad Jizerou
  - Nemocnice Kyjov, prispevkova organizace, Infekcni oddeleni, Kyjov
  - Slezska Nemocnice v Opave, prispevkova organizace, Opava
  - Policska nemocnice s.r.o.,, Polička
  - Fakultni nemocnice v Motole, Prague
  - Oblastni nemocnice Pribram, a.s., Pribram I.
  - Interna a kardiologie s.r.o., Rožnov pod Radhoštěm
  - Nemocnice Slany, p.o., Slaný
  - Sarkamed s.r.o., Slaný
  - Krajska zdravotni, a.s., Masarykova nemocnice Usti nad Labem, Ústí nad Labem
- Finland (6):
  - Helsinki University Central Hospital, Helsinki
  - Kokkola Vaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- France (4):
  - CHU DIJON BOURGOGNE- Hopital Francois Mitterrand, Dijon
  - CIC Vaccinologie Cochin- Pasteur 1417, Paris
  - Hopital Nord-CHU Saint Etienne, Saint-Priest-en-Jarez
  - CHRU de Tours- Hopital Bretonneau, Tours
- Germany (11):
  - Emovis GmbH, Berlin
  - MECS Cottbus GmbH, Cottbus
  - Diabetologische Gemeinschaftspraxis Dr. Schaper & Dr. Faulmann, Dresden
  - Universitaetsklinikum Essen, Klinik fuer Infektiologie, Essen
  - EUGASTRO GmbH/ Praxis, Leipzig
  - SIBAmed Studienzentrum GmbH & Co.KG, Leipzig
  - Gemeinschaftspraxis Dr. med. Heidrun Taeschner und Dr. med. Susanne Bonigut, Leipzig
  - Universitaetsmedizin Rostock, Rostock
  - Praxis Dr. med. J. Springub/ W. Schwarz, Westerstede
  - Studienzentrum Nordwest, Westerstede
  - Klinikum Wuerzburg Mitte gGmbH, Würzburg
- Hungary (9):
  - Bajai Szent Rokus Korhaz, II Belgyogyaszat, Baja
  - DRC Kft., Balatonfüred
  - Budapesti Szent Ferenc Korhaz, Kardiologiai Rehabilitacios Osztaly, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, I. Belgyogyaszati Osztaly, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, VI. Osztaly, Budapest
  - Semmelweis Egyetem III. Sz. Belgyogyaszati Klinika, Budapest
  - ClinTrial Audit Kft., Klinikai Farmakologiai Intezet, Vedooltasi Ambulancia, Debrecen
  - CRU Hungary Kft., Encs
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Infektologiai Osztaly, Kaposvár
- Japan (25):
  - Tokai Memorial Hospital, Kasugai, Aichi-ken
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Daido Clinic, Nagoya, Aichi-ken
  - Kamiiida daiichi General Hospital, Nagoya, Aichi-ken
  - Iizuka Hospital, Iizuka, Fukuoka
  - Seishinkai Inoue Hospital, Itoshima, Fukuoka
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Kenwakai Otemachi Hospital, Kitakyushu, Fukuoka
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Miyanomori Memorial Hospital, Sapporo, Hokkaido
  - Medical Corporation Tokushukai Koga General Hospital, Koga, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Osaki Citizen Hospital, Ōsaki, Miyagi
  - Social Medical Care Corporation Hose-kai Marunouchi Hospital, Matsumoto, Nagano
  - Nozaki Tokushukai Hospital, Daitō, Osaka
  - Omi Medical Center, Kusatsu, Shiga
  - Yaizu City Hospital, Yaizu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Nerima General Hospital, Nerima-ku, Tokyo
  - Sekino Hospital, Toshima-ku, Tokyo
  - Fukui-Ken Saiseikai Hospital, Fukui
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Saga-Ken Medical Centre Koseikan, Saga
- Peru (4):
  - Hospital Cayetano Heredia, San Martín de Porres, Lima region
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Clinica Internacional S.A, Lima
  - Centro de Investigaciones Biomédicas - CIBIOM/Clinica Peruano Americana S.A, Trujillo, La Libertad
- Poland (8):
  - NZOZ Vitamed, Bydgoszcz
  - Synexus Polska Sp. z o.o Oddzial w Gdansku, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - SYNEXUS Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Synexus Polska Sp. z o.o. Oddział w Poznaniu, Poznan
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Salmed S. C., Łęczna
- Portugal (5):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar do Baixo Vouga, E.P.E., Aveiro
  - Hospital de Braga, Braga
  - Hospital Senhora de Oliveira - Guimaraes, E.P.E., Guimarães
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Slovakia (13):
  - PULMO-MEDIK s.r.o., Pneumologicko-ftizeologicka ambulancia, Bojnice
  - Medak s.r.o., Gastroenterologicka ambulancia, Bratislava
  - Stalerg, s.r.o., Košice
  - KM Management spol. s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Dionea, s.r.o., Nové Zámky
  - MEDIPA, s.r.o., Piešťany
  - MUDr. Viliam Cibik, PhD, s.r.o., Pruské
  - Medilex s.r.o., Interna ambulancia, Rimavská Sobota
  - Plucna ambulancia Hrebenar s.r.o., Spišská Nová Ves
  - SPAOLO s.r.o., Ambulancia vnutorneho lekarstva, Stará Turá
  - Privatna urologicka ambulancia, s.r.o., Trenčín
  - MUDr. Zakova, s.r.o., Trenčín
  - Fakutna nemocnica Trnava, Trnava
- South Korea (13):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Asan Medical Center, Songpa-gu, Seoul
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (12):
  - EAP Centelles, Centelles, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Parc de Salut Mar- Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (5):
  - Infektionskliniken, Malarsjukhuset, Eskilstuna
  - Gothia Forum CTC/Sahlgrenska Universitetssjukhuset, Gothenburg
  - Sahlgrenska Universitetssjukhuset - Ostra Sjukhuset, Gothenburg
  - Avdelningen for kliniska provningar, S-huset, Örebro
  - Karolinska Trial Alliance, KTA Prim Sabbatsbergs sjukhus, Stockholm
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan (r.o.c.)
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
- United Kingdom (13):
  - Stockport Nhs Foundation Trust, Stockport, Cheshire
  - Fowey River Practice, Fowey, Cornwall
  - Oak Tree Surgery, Liskeard, Cornwall
  - The Alverton Practise, St Clare Medical Centre, Penzance, Cornwall
  - Rame Group Practice, Rame Medical Ltd., Torpoint, Cornwall
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Knowle House Surgery, Plymouth, Devon
  - Layton Medical Centre, Blackpool, Lancashire
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - NHS Lothian, Western General Hospital, Edinburgh, Midlothian
  - Heart of England NHS Foundation Trust, Birmingham, WEST Midlands
  - St James University Hospital, Leeds
  - Newcastle upon Tyne Hospitals NHS Foundation trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Donskey CJ, Dubberke ER, Klein NP, Liles EG, Szymkowiak K, Wilcox MH, Lawrence J, Bouguermouh S, Zhang H, Koury K, Bailey R, Smith HM, Lockhart S, Lamberth E, Kalina WV, Pride MW, Webber C, Anderson AS, Jansen KU, Gruber WC, Kitchin N. CLOVER (CLOstridium difficile Vaccine Efficacy tRial) Study: A Phase 3, Randomized Trial Investigating the Efficacy and Safety of a Detoxified Toxin A/B Vaccine in Adults 50 Years and Older at Increased Risk of Clostridioides difficile Infection. Clin Infect Dis. 2024 Dec 17;79(6):1503-1511. doi: 10.1093/cid/ciae410. PMID 39180325
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5091007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18095 participants signed the informed consent form (ICF). Among that 560 participants did not meet all eligibility criteria, were not randomized and vaccinated. Overall, 17535 participants were randomized, out of which only 17440 participants received at least 1 dose of the investigational product.
Groups:
- Clostridium Difficile Vaccine: Participants were randomized to Clostridium difficile vaccine 200 microgram total toxoid per dose intramuscularly at Months 0, 1 and 6.
- Placebo: Participants were randomized to placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly at Months 0, 1 and 6.
Period: Overall Study
Arm/Group | Clostridium Difficile Vaccine | Placebo
Started | 8766 | 8769
Vaccinated at Month 0 (Dose 1) (Among 8766 participants randomized to Clostridium difficile vaccine(Cdif.vac)group(grp),8723 received first dose, 8769 randomized to placebo grp,8717 received first dose. But 2 participants in Cdif.vac grp received placebo,1 participant in placebo grp received Cdif.vac for first dose.So, 8722 received Cdif.vac, 8718 received placebo for first dose. 8722 and 8718=participants in baseline characteristics, safety data summaries since safety population based on actual vaccine received at first dose.) | 8723 | 8717
Received Clostridium Difficile Vaccine | 8721 | 1
Received Placebo | 2 | 8716
Vaccinated at Month 1 (Dose 2) | 8311 | 8331
Received Clostridium Difficile Vaccine | 8310 | 0
Received Placebo | 1 | 8331
Vaccinated at Month 6 (Dose 3) | 7894 | 7967
Received Clostridium Difficile Vaccine | 7894 | 0
Received Placebo | 0 | 7967
Completed | 5533 | 5574
Not Completed | 3233 | 3195
Not completed — Adverse Event | 90 | 72
Not completed — Death | 365 | 358
Not completed — Lost to Follow-up | 382 | 394
Not completed — Physician Decision | 77 | 66
Not completed — Protocol Violation | 43 | 52
Not completed — Withdrawal by Subject | 2160 | 2133
Not completed — Site terminated | 7 | 8
Not completed — Other | 66 | 60
Not completed — Withdrawn before any study vaccination | 43 | 52

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product.
Groups:
- Clostridium Difficile Vaccine: Participants who received Clostridium difficile vaccine 200 microgram total toxoid per dose intramuscularly at Months 0, 1 and 6.
- Placebo: Participants who received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly at Months 0, 1 and 6.
- Total: Total of all reporting groups
Arm/Group | Clostridium Difficile Vaccine | Placebo | Total
Number analyzed (Participants) | 8722 | 8718 | 17440
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.5) | 68.1 (7.5) | 68.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4472 | 4501 | 8973
  Male | 4250 | 4217 | 8467
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1119 | 1143 | 2262
  Not Hispanic or Latino | 7546 | 7515 | 15061
  Unknown or Not Reported | 57 | 60 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 53 | 54 | 107
  Asian | 754 | 725 | 1479
  Native Hawaiian or Other Pacific Islander | 20 | 14 | 34
  Black or African American | 663 | 666 | 1329
  White | 6891 | 6922 | 13813
  More than one race | 327 | 322 | 649
  Unknown or Not Reported | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of First Primary Episodes of Clostridium Difficile Infection (CDI) (Definition 1) Follow-up After Dose 3
Description: CDI definition 1 for a primary episode of CDI (no previous CDI onset in the prior 8 weeks) was defined as either a) presence of diarrhea, defined as passage of 3 or more unformed stools (Bristol stool chart types 5-7) in 24 or fewer consecutive hours, and stool sample that was positive for the toxin B gene (by polymerase chain reaction [PCR)] and positive for toxin A and/or toxin B, as measured in the central laboratory; or b) Pseudomembranous colitis diagnosed at colonoscopy, at surgery, or histopathologically; and corresponding stool sample that was positive for the toxin B gene (via PCR) as measured in the central laboratory. End of surveillance period was defined as accumulation of at least 40 CDI cases.
Time Frame: From 14 days after Dose 3 to the end of the surveillance period (mean follow-up after dose 3 was 34.2 months)
Population: Per Protocol-3 analysis population included all randomized participants who received dose 1, dose 2, and dose 3 of the investigational product to which they were randomized and had no major protocol violations up to and including 14 days after dose 3. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Episodes
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 7707 | 7805
Episodes | 17 | 25
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority — Lower bound of confidence interval greater than 20% demonstrate vaccine efficacy; Vaccine efficacy = 31.0, 96.4% CI 2-sided [-38.7 to 66.6] — Vaccine efficacy(VE)=100*(1-infection rate ratio[IRR]),IRR=calculated ratio of first primary CDI incidence between Clostridium difficile vaccine group and placebo group. 96.4% CI was estimated using Clopper-Pearson-Method

2. Primary Outcome: Number of First Primary Episodes of Clostridium Difficile Infection (CDI) (Definition 1) Follow-up After Dose 2
Description: CDI definition 1 for a primary episode of CDI (no previous CDI onset in the prior 8 weeks) was defined as either a) presence of diarrhea, defined as passage of 3 or more unformed stools (Bristol stool chart types 5-7) in 24 or fewer consecutive hours, and stool sample that was positive for the toxin B gene (by PCR) and positive for toxin A and/or toxin B, as measured in the central laboratory; or b) Pseudomembranous colitis diagnosed at colonoscopy, at surgery, or histopathologically; and corresponding stool sample that was positive for the toxin B gene (via PCR) as measured in the central laboratory. End of surveillance period was defined as accumulation of at least 40 CDI cases.
Time Frame: From 14 days after Dose 2 to the end of the surveillance period (mean follow-up after dose 2 was 36 months)
Population: Per Protocol-2 analysis population included all randomized participants who received dose 1 and dose 2 of the investigational product to which they were randomized and had no major protocol violations up to and including 14 days after dose 2. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Episodes
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8139 | 8184
Episodes | 24 | 34
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority — Lower bound of confidence interval greater than 20% demonstrate vaccine efficacy; Vaccine efficacy = 28.6, 96.4% CI 2-sided [-28.4 to 61.0] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Dose 1
Description: Local reactions included redness, swelling and pain at injection site. These were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. One measuring device unit= 0.5 centimeter (cm) and graded as mild: 2.5 to 5.0 cm, moderate: greater than (>) 5.0 to 10.0 cm, severe: >10.0 cm. Grade 4 indicated necrosis or exfoliative dermatitis for redness and necrosis for swelling Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity. Grade 4 indicated emergency room visit or hospitalization.
Time Frame: Within 7 days after Dose 1 at Month 0
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8558 | 8510
Percentage of participants
  Redness: Mild | 1.5 [1.3 to 1.8] | 0.6 [0.4 to 0.7]
  Redness: Moderate | 0.5 [0.4 to 0.7] | 0.3 [0.2 to 0.4]
  Redness: Severe | 0.4 [0.3 to 0.6] | 0.2 [0.1 to 0.3]
  Redness: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Swelling: Mild | 1.5 [1.3 to 1.8] | 0.5 [0.3 to 0.7]
  Swelling: Moderate | 0.9 [0.8 to 1.2] | 0.3 [0.2 to 0.5]
  Swelling: Severe | 0.3 [0.2 to 0.5] | 0.1 [0.0 to 0.2]
  Swelling: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Pain at injection site: Mild | 17.5 [16.7 to 18.3] | 6.2 [5.7 to 6.8]
  Pain at injection site: Moderate | 2.2 [1.9 to 2.5] | 0.8 [0.6 to 1.0]
  Pain at injection site: Severe | 0.1 [0.0 to 0.2] | 0.1 [0.1 to 0.2]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.0] | 0.1 [0.0 to 0.1]

4. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Dose 2
Description: Local reactions included redness, swelling and pain at injection site. These were recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. One measuring device unit= 0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm, severe: >10.0 cm. Grade 4 indicated necrosis or exfoliative dermatitis for redness and necrosis for swelling. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity. Grade 4 indicated emergency room visit or hospitalization.
Time Frame: Within 7 days after Dose 2 at Month 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8041 | 8039
Percentage of participants
  Redness: Mild | 2.6 [2.2 to 2.9] | 0.3 [0.2 to 0.5]
  Redness: Moderate | 2.2 [1.9 to 2.6] | 0.2 [0.1 to 0.3]
  Redness: Severe | 0.9 [0.7 to 1.2] | 0.1 [0.0 to 0.1]
  Redness: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Swelling: Mild | 3.2 [2.8 to 3.6] | 0.3 [0.2 to 0.5]
  Swelling: Moderate | 3.0 [2.6 to 3.4] | 0.2 [0.1 to 0.3]
  Swelling: Severe | 0.9 [0.7 to 1.1] | 0.1 [0.0 to 0.2]
  Swelling: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Pain at injection site: Mild | 23.0 [22.1 to 23.9] | 4.3 [3.9 to 4.8]
  Pain at injection site: Moderate | 4.5 [4.0 to 4.9] | 0.7 [0.5 to 0.9]
  Pain at injection site: Severe | 0.2 [0.1 to 0.3] | 0.1 [0.0 to 0.1]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

5. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Dose 3
Description: as for outcome 4
Time Frame: Within 7 days after Dose 3 at Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 7526 | 7569
Percentage of participants
  Redness: Mild | 2.6 [2.3 to 3.0] | 0.4 [0.2 to 0.5]
  Redness: Moderate | 2.4 [2.1 to 2.8] | 0.2 [0.1 to 0.4]
  Redness: Severe | 0.7 [0.5 to 0.9] | 0.1 [0.0 to 0.1]
  Redness: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Swelling: Mild | 3.5 [3.1 to 3.9] | 0.3 [0.2 to 0.5]
  Swelling: Moderate | 3.3 [2.9 to 3.7] | 0.2 [0.1 to 0.4]
  Swelling: Severe | 0.8 [0.6 to 1.1] | 0 [0.0 to 0.0]
  Swelling: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Pain at injection site: Mild | 21.0 [20.1 to 21.9] | 3.6 [3.2 to 4.1]
  Pain at injection site: Moderate | 4.5 [4.0 to 5.0] | 0.8 [0.6 to 1.0]
  Pain at injection site: Severe | 0.2 [0.1 to 0.4] | 0.1 [0.0 to 0.1]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Dose 1
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild: (38.0 to 38.4 degree Celsius [deg C]), moderate: (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C), potentially life threatening (> 40.0 deg C). Fatigue, headache, joint pain and muscle pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration, grade 4: emergency room visit or hospitalization for hypotensive shock.
Time Frame: Within 7 days after Dose 1 at Month 0
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8558 | 8510
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.5 [0.3 to 0.6] | 0.4 [0.3 to 0.5]
  Fever: 38.5-38.9 deg C | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  Fever: 39.0-40.0 deg C | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  Fever: >40.0 deg C | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.2]
  Fatigue: Mild | 11.6 [10.9 to 12.3] | 10.2 [9.6 to 10.9]
  Fatigue: Moderate | 10.6 [10.0 to 11.3] | 10.4 [9.7 to 11.0]
  Fatigue: Severe | 1.1 [0.9 to 1.3] | 1.2 [1.0 to 1.5]
  Fatigue: Grade 4 | 0.1 [0.0 to 0.1] | 0 [0.0 to 0.0]
  Headache: Mild | 11.6 [10.9 to 12.3] | 10.1 [9.4 to 10.7]
  Headache: Moderate | 5.8 [5.3 to 6.3] | 5.4 [4.9 to 5.9]
  Headache: Severe | 0.5 [0.4 to 0.7] | 0.6 [0.5 to 0.8]
  Headache: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Vomiting: Mild | 1.1 [0.8 to 1.3] | 0.7 [0.5 to 0.9]
  Vomiting: Moderate | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3]
  Vomiting: Severe | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Vomiting: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  New or worsening muscle pain: Mild | 5.2 [4.7 to 5.7] | 3.9 [3.5 to 4.3]
  New or worsening muscle pain: Moderate | 5.7 [5.2 to 6.2] | 5.6 [5.1 to 6.1]
  New or worsening muscle pain: Severe | 0.6 [0.4 to 0.8] | 0.6 [0.5 to 0.8]
  New or worsening muscle pain: Grade 4 | 0.1 [0.0 to 0.1] | 0 [0.0 to 0.0]
  New or worsening joint pain: Mild | 4.0 [3.6 to 4.5] | 3.3 [2.9 to 3.7]
  New or worsening joint pain: Moderate | 5.2 [4.7 to 5.7] | 5.0 [4.5 to 5.5]
  New or worsening joint pain: Severe | 0.5 [0.4 to 0.7] | 0.5 [0.3 to 0.6]
  New or worsening joint pain: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Dose 2
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild: (38.0 to 38.4 deg C), moderate: (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C), potentially life threatening (> 40.0 deg C). Fatigue, headache, joint pain and muscle pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration, grade 4: emergency room visit or hospitalization for hypotensive shock.
Time Frame: Within 7 days after Dose 2 at Month 1
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''number analyzed'' signifies number of participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8041 | 8039
Percentage of participants
  Fever: 38.0-38.4 deg C: number analyzed (Participants) | 8041 | 8038
  Fever: 38.0-38.4 deg C | 0.4 [0.3 to 0.6] | 0.4 [0.3 to 0.6]
  Fever: 38.5-38.9 deg C: number analyzed (Participants) | 8041 | 8038
  Fever: 38.5-38.9 deg C | 0.2 [0.1 to 0.3] | 0.1 [0.0 to 0.2]
  Fever: 39.0-40.0 deg C: number analyzed (Participants) | 8041 | 8038
  Fever: 39.0-40.0 deg C | 0.1 [0.0 to 0.2] | 0.2 [0.1 to 0.3]
  Fever: >40.0 deg C: number analyzed (Participants) | 8041 | 8038
  Fever: >40.0 deg C | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Fatigue: Mild | 10.2 [9.6 to 10.9] | 7.8 [7.2 to 8.4]
  Fatigue: Moderate | 9.4 [8.7 to 10.0] | 9.0 [8.4 to 9.6]
  Fatigue: Severe | 1.0 [0.8 to 1.2] | 1.0 [0.8 to 1.2]
  Fatigue: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Headache: Mild | 10.1 [9.4 to 10.8] | 8.3 [7.7 to 9.0]
  Headache: Moderate | 5.1 [4.6 to 5.6] | 5.5 [5.0 to 6.1]
  Headache: Severe | 0.5 [0.4 to 0.7] | 0.4 [0.3 to 0.6]
  Headache: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Vomiting: Mild | 0.8 [0.6 to 1.0] | 0.7 [0.5 to 0.9]
  Vomiting: Moderate | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3]
  Vomiting: Severe | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Vomiting: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  New or worsening muscle pain: Mild | 4.8 [4.3 to 5.3] | 3.2 [2.9 to 3.6]
  New or worsening muscle pain: Moderate | 5.1 [4.6 to 5.6] | 4.2 [3.8 to 4.7]
  New or worsening muscle pain: Severe | 0.5 [0.4 to 0.7] | 0.6 [0.4 to 0.8]
  New or worsening muscle pain: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  New or worsening joint pain: Mild | 3.8 [3.4 to 4.2] | 2.9 [2.6 to 3.3]
  New or worsening joint pain: Moderate | 4.6 [4.1 to 5.0] | 3.9 [3.5 to 4.4]
  New or worsening joint pain: Severe | 0.4 [0.3 to 0.6] | 0.5 [0.3 to 0.6]
  New or worsening joint pain: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

8. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Dose 3
Description: as for outcome 7
Time Frame: Within 7 days after Dose 3 at Month 6
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 7526 | 7569
Percentage of participants
  Fever: 38.0-38.4 deg C: number analyzed (Participants) | 7525 | 7569
  Fever: 38.0-38.4 deg C | 0.4 [0.3 to 0.6] | 0.2 [0.1 to 0.4]
  Fever: 38.5-38.9 deg C: number analyzed (Participants) | 7525 | 7569
  Fever: 38.5-38.9 deg C | 0.1 [0.1 to 0.2] | 0.1 [0.0 to 0.2]
  Fever: 39.0-40.0 deg C: number analyzed (Participants) | 7525 | 7569
  Fever: 39.0-40.0 deg C | 0.1 [0.1 to 0.2] | 0.1 [0.0 to 0.2]
  Fever: >40.0 deg C: number analyzed (Participants) | 7525 | 7569
  Fever: >40.0 deg C | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Fatigue: Mild | 9.2 [8.6 to 9.9] | 7.0 [6.4 to 7.6]
  Fatigue: Moderate | 9.4 [8.7 to 10.0] | 8.0 [7.4 to 8.6]
  Fatigue: Severe | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0]
  Fatigue: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Headache: Mild | 8.4 [7.8 to 9.0] | 7.9 [7.3 to 8.5]
  Headache: Moderate | 5.7 [5.1 to 6.2] | 4.7 [4.2 to 5.2]
  Headache: Severe | 0.3 [0.2 to 0.5] | 0.5 [0.3 to 0.6]
  Headache: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Vomiting: Mild | 0.6 [0.5 to 0.8] | 0.5 [0.4 to 0.7]
  Vomiting: Moderate | 0.1 [0.0 to 0.2] | 0.2 [0.1 to 0.3]
  Vomiting: Severe | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Vomiting: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  New or worsening muscle pain: Mild | 4.0 [3.5 to 4.4] | 2.5 [2.2 to 2.9]
  New or worsening muscle pain: Moderate | 4.8 [4.3 to 5.3] | 4.1 [3.6 to 4.6]
  New or worsening muscle pain: Severe | 0.5 [0.3 to 0.7] | 0.5 [0.3 to 0.7]
  New or worsening muscle pain: Grade 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  New or worsening joint pain: Mild | 3.0 [2.6 to 3.4] | 2.5 [2.2 to 2.9]
  New or worsening joint pain: Moderate | 4.4 [3.9 to 4.8] | 3.6 [3.2 to 4.0]
  New or worsening joint pain: Severe | 0.4 [0.3 to 0.6] | 0.4 [0.3 to 0.5]
  New or worsening joint pain: Grade 4 | 0.1 [0.0 to 0.1] | 0 [0.0 to 0.0]

9. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and all non-serious adverse events. An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event. AEs included both SAEs and all Non-SAEs (except local and systemic events).
Time Frame: From Day 1 of Dose 1 to 1 Month after Dose 3 (7 Months)
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8722 | 8718
Participants
  Any AEs | 4161 | 4050
  Non-Serious AEs | 3913 | 3791

10. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: From Day 1 of Dose 1 up to 6 months after Dose 3 (up to Month 12)
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8722 | 8718
Participants | 719 | 722

11. Secondary Outcome: Number of All Episodes of CDI (Definition 1 and 2) After Dose 3
Description: CDI definition 1 for primary episode of CDI (no previous CDI onset in prior 8 weeks) and CDI definition 2 for recurrent episode (episode occurred 8 weeks or less after onset of previous episode [provided symptoms of previous episode resolved]) were both defined as either a) presence of diarrhea, (passage of 3 or more unformed stools [Bristol stool chart types 5-7]) in 24 or fewer consecutive hours, stool sample positive for toxin B gene (by PCR),positive for toxin A and/or toxin B, as measured in central laboratory; or b) Pseudomembranous colitis diagnosed at colonoscopy, surgery, histopathologically; and corresponding stool sample positive for toxin B gene (via PCR) as measured in central laboratory. End of surveillance period was defined as accumulation of at least 40 CDI cases.
Time Frame: From 14 days after Dose 3 to the end of the surveillance period (mean follow-up after dose 3 was 34.2 months)
Population: as for outcome 1
Measure: Number; unit: Episodes
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 7707 | 7805
Episodes | 28 | 32
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Vaccine efficacy = 11.1, 98.2% CI 2-sided [-110.7 to 62.5] — VE = 100*(1 - Hazard Ratio). 98.2% CI was estimated using Proportional Means Model

12. Secondary Outcome: Time to Resolution for Participants With First Primary Episodes of CDI (Definition 1) After Dose 3
Description: Resolution of the event was the last day on which the event was recorded in the e-diary or the date the event ends if it was unresolved during the participant diary-recording period (end date collected on the case report form [CRF]). CDI definition 1 for a primary episode of CDI (no previous CDI onset in the prior 8 weeks) was defined as either a) presence of diarrhea, defined as passage of 3 or more unformed stools (Bristol stool chart types 5-7) in 24 or fewer consecutive hours, and stool sample that was positive for the toxin B gene (by PCR) and positive for toxin A and/or toxin B, as measured in the central laboratory; or b) Pseudomembranous colitis diagnosed at colonoscopy, at surgery, or histopathologically; and corresponding stool sample that was positive for the toxin B gene (via PCR) as measured in the central laboratory. End of surveillance period was defined as accumulation of at least 40 CDI cases.
Time Frame: From 14 days after Dose 3 to the end of the surveillance period (mean follow-up after dose 3 was 34.2 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 17 | 24
Days | 1.0 [1 to 18] | 4.0 [1 to 183]
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; p = 0.0172, Wilcoxon Rank Sum Test (2-sided)

13. Secondary Outcome: Proportion of Participants Who Required Medical Attention During First Primary Episode of CDI (Definition 1) After Dose 3
Description: as for outcome 2
Time Frame: From 14 days after Dose 3 to the end of the surveillance period (mean follow-up after dose 3 was 34.2 months)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 17 | 25
Proportion of participants | 0 | 0.440
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Ratio of proportions = 0.000, 98.2% CI 2-sided [0.00 to 0.81]

14. Secondary Outcome: Number of Participants With Recurrent Episodes of CDI (Definition 2) After Dose 3
Description: CDI definition 2 for a recurrent episode (an episode of CDI that occurred 8 weeks or less after the onset of a previous CDI episode [provided the symptoms of the previous episode had resolved]), was defined as either a) presence of diarrhea, defined as passage of 3 or more unformed stools (Bristol stool chart types 5-7) in 24 or fewer consecutive hours; and stool sample that was positive for the toxin B gene (by PCR) and positive for toxin A and/or toxin B, as measured in the central laboratory; or b) Pseudomembranous colitis diagnosed at colonoscopy, at surgery, or histopathologically; and corresponding stool sample that was positive for the toxin B gene (by PCR) as measured in the central laboratory. End of surveillance period was defined as accumulation of at least 40 CDI cases.
Time Frame: From 14 days after Dose 3 to the end of the surveillance period (mean follow-up after dose 3 was 34.2 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 7707 | 7805
Participants | 5 | 3
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Vaccine efficacy = -69.3, 98.2% CI 2-sided [-1533.1 to 75.6] — Vaccine efficacy(VE)=100*(1-infection rate ratio[IRR]),IRR=calculated ratio of recurrent CDI incidence between Clostridium difficile vaccine group and placebo group. 98.2% CI was estimated using Clopper-Pearson-Method

15. Secondary Outcome: Number of All Episodes of CDI (Definition 1 and 2) After Dose 2
Description: as for outcome 11
Time Frame: From 14 days after Dose 2 to the end of the surveillance period (mean follow-up after dose 2 was 36 months)
Population: as for outcome 2
Measure: Number; unit: Episodes
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8139 | 8184
Episodes | 37 | 44
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Vaccine efficacy = 14.9, 98.2% CI 2-sided [-74.6 to 58.5] — VE = 100*(1 - Hazard Ratio). 98.2% CI was estimated using Proportional Means Model

16. Secondary Outcome: Number of Participants With Recurrent Episodes of CDI (Definition 2) After Dose 2
Description: as for outcome 14
Time Frame: From 14 days after Dose 2 to the end of the surveillance period (mean follow-up after dose 2 was 36 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8139 | 8184
Participants | 6 | 3
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Vaccine efficacy = -102.4, 98.2% CI 2-sided [-1770.1 to 67.2] — VE = 100*(1 - IRR), where IRR= the calculated ratio of recurrent CDI incidence between the Clostridium difficile vaccine group and the placebo group. 98.2% CI was estimated using Clopper-Pearson-Method

17. Secondary Outcome: Number of First Primary Episode of CDI (Definition 1) After Dose 2 and Before Dose 3
Description: as for outcome 2
Time Frame: From 14 days after Dose 2 to Dose 3 or the day the third vaccination was expected (168 days after Dose 2) for participants who received only 2 doses
Population: as for outcome 2
Measure: Number; unit: Episodes
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8139 | 8184
Episodes | 7 | 8
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine vs Placebo; Test type: Superiority; Vaccine efficacy = 12.0, 98.2% CI 2-sided [-246.7 to 78.5] — Vaccine efficacy(VE)=100*(1-infection rate ratio[IRR]),IRR=calculated ratio of first primary CDI incidence between Clostridium difficile vaccine group and placebo group. 98.2% CI was estimated using Clopper-Pearson-Method

18. Secondary Outcome: Number of Participants With Recurrent Episode of CDI (Definition 2) After Dose 2 and Before Dose 3
Description: as for outcome 14
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clostridium Difficile Vaccine | Placebo
Number analyzed (Participants) | 8139 | 8184
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (included in other AEs): within 7 days after each dose (systematic assessment); SAEs: from Day 1 up to 6 months after last dose of vaccination (up to 12 months); other AEs: from Day 1 up to 1 month after last dose of vaccination (up to 7 months); All-Cause mortality: from Day 1 up to 6 months after last dose of vaccination (up to 12 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Cause of death was unknown. Safety analysis population included all participants who received at least 1 dose of the investigational product.
Arm/Group | Clostridium Difficile Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 369/8722 | 362/8718
Serious Adverse Events (participants affected / at risk) | 719/8722 | 722/8718
Other Adverse Events (participants affected / at risk) | 5702/8722 | 4314/8718
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clostridium Difficile Vaccine (N=8722) | Placebo (N=8718)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 20 | 8
Angina pectoris (Cardiac disorders) | 9 | 13
Angina unstable (Cardiac disorders) | 4 | 9
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 12 | 15
Atrial flutter (Cardiac disorders) | 4 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 3 | 3
Cardiac arrest (Cardiac disorders) | 3 | 6
Cardiac failure acute (Cardiac disorders) | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 14 | 17
Cardiac failure (Cardiac disorders) | 13 | 10
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 3 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 13 | 8
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 5
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 12 | 4
Myocardial injury (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 4
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 3 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 3
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Hereditary motor and sensory neuropathy (Congenital, familial and genetic disorders) | 0 | 1
Mobile caecum syndrome (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3
Basedow's disease (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 4
Epiretinal membrane (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 2
Retinal vein occlusion (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 6
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Anastomotic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 2 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 3
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 8 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 4
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Adverse drug reaction (General disorders) | 0 | 2
Asthenia (General disorders) | 6 | 3
Chest discomfort (General disorders) | 1 | 2
Chest pain (General disorders) | 25 | 32
Complication of device insertion (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Drug interaction (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 3
Injection site haematoma (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 3 | 0
Pacemaker generated arrhythmia (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 1 | 0
Surgical failure (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 3 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 5
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 3
Abscess neck (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 5
Arthritis bacterial (Infections and infestations) | 3 | 2
Arthritis infective (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 12 | 11
Bursitis infective (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 23 | 18
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 3
Cystitis escherichia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 2 | 3
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 8 | 7
Empyema (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fournier's gangrene (Infections and infestations) | 1 | 0
Fracture infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 2
Gas gangrene (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 5
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Haemorrhagic fever with renal syndrome (Infections and infestations) | 0 | 1
Haemorrhagic fever (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 2
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 6 | 4
Intervertebral discitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Listeria sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 5 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 0 | 1
Medical device site joint infection (Infections and infestations) | 2 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 2 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 2 | 0
Osteomyelitis fungal (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 12 | 11
Parotitis (Infections and infestations) | 1 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 3
Pneumonia bacterial (Infections and infestations) | 2 | 2
Pneumonia influenzal (Infections and infestations) | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 38 | 39
Post procedural infection (Infections and infestations) | 3 | 0
Postoperative wound infection (Infections and infestations) | 2 | 1
Prostate infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 3
Pyelonephritis (Infections and infestations) | 2 | 2
Pyuria (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 16 | 16
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 3 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 13 | 10
Urosepsis (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 4
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Combined tibia-fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 10
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 7
Femur fracture (Injury, poisoning and procedural complications) | 2 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 5
Incision site swelling (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 2
Intentional product misuse (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 6 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 2 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Postpolypectomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 4
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 5
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypoosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 9
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 2
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 1
Synovial disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell small lymphocytic lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 2 | 1
Brain injury (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 11 | 7
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 2 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2
Encephalopathy (Nervous system disorders) | 4 | 3
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 6 | 5
Lacunar infarction (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 3 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Occipital neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 2
Spinal stroke (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 11 | 13
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 8 | 2
Wernicke-Korsakoff syndrome (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 3
Device loosening (Product Issues) | 1 | 2
Device occlusion (Product Issues) | 1 | 0
Lead dislodgement (Product Issues) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 2
Depression suicidal (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 4
Major depression (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Paranoia (Psychiatric disorders) | 1 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 9 | 18
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Contracted bladder (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Incontinence (Renal and urinary disorders) | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 3
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Subcapsular renal haematoma (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 2
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 3
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 2 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 33 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Cellulite (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 3
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Physical assault (Social circumstances) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 3 | 3
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 7
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypertensive crisis (Vascular disorders) | 3 | 1
Hypertensive emergency (Vascular disorders) | 5 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 8
Iliac artery occlusion (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 2
Subclavian steal syndrome (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Vein disorder (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clostridium Difficile Vaccine (N=8722) | Placebo (N=8718)
Fatigue (FATIGUE) (General disorders) | 3240 | 2820
Injection site erythema (REDNESS) (General disorders) | 1879 | 653
Injection site pain (PAIN) (General disorders) | 3596 | 1056
Injection site swelling (SWELLING) (General disorders) | 1846 | 414
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 1583 | 1354
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 1856 | 1487
Headache (HEADACHE) (Nervous system disorders) | 2615 | 2323

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03090191/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT03090191/SAP_001.pdf